CLINICAL TRIAL: NCT03974997
Title: TNF-related Weak Inducer of Apoptosis (TWEAK), a New Biomarker Predicting Inflammatory Thrust in Multiple Sclerosis
Brief Title: Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019-12
Record Dates: First submitted 2019-06-03; First posted 2019-06-05 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: This is a single-center interventional study with minimal risks and constraints on a cohort of MS patients. Patients with clinically isolated syndrome suggestive of MS will be included prospectively and consecutively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- serum concentration changes in cytokine TWEAK (Other): We will perform a prospective study in which 50 patients with multiple sclerosis in the isolated clinical syndrome stage will be included over a 12-month period. Mental Cerebral MRIs will be performed for each patient at baseline (T0), month 6, and month 12. Serum dosages of TWEAK will be performed each month for each patient for one year. Patients will also be treated with soluble TNF, the leader in the TNF family of ligands, anti-TWEAK antibodies (which may interfere with the activity and dosage of TWEAK) as well as C-reactive Protein C ( search for intercurrent infectious episode). These dosages will be correlated with the clinical evolution (appearance or not of an inflammatory flare) as well as the data of the imagery (number of lesions raised or not by the gadolinium).
  Interventions: Diagnostic Test: Determination of the circulating serum concentration of cytoquine TWEAK

INTERVENTIONS:
Diagnostic Test: Determination of the circulating serum concentration of cytoquine TWEAK — Blood samples (20 ml of blood on dry tube) by venipuncture at the bend of the elbow will be made at T0, then monthly for a period of 1 year . The sera will be isolated by centrifugation and then frozen at -80 degrees Assays of the soluble form of TWEAK and TNF will be performed by ELISA blot technique developed by the team.

SUMMARY:
A significant variation in the serum concentration of the circulating cytokine TWEAK is associated with the onset of an inflammatory attack of MS. Study the concentration variations of the serum soluble form of cytokine TWEAK during the first year of MS and to analyze their correlation with the occurrence of an inflammatory disease outbreak.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is the most common chronic autoimmune demyelinating and neurodegenerative disease of the central nervous system (CNS) of disabling neurological diseases in young adults in France. Patients with MS can present a wide range of symptoms spread over time and space such as motor, sensory, visual or vesico-sphincter deficits. One of the current challenges in treating patients with symptoms suggestive of MS is to assess the risk of an inflammatory flare in order to avoid or limit the installation of an irreversible neurological handicap. At present, the inflammatory activity of the disease is evaluable only by cerebral imaging (MRI). However, these examinations can not be carried out as often as necessary because of their accessibility, cost, duration and the potential deleterious effects of gadolinium accumulation. This is why a blood biomarker able to report early on the inflammatory activity of the disease would be of great help during the monitoring and treatment of patients. TWEAK (TNF-related weak inducer of apoptosis or TNFSF12) is a pro-inflammatory cytokine member of the TNF family. This cytokine is overexpressed in tissues with chronic inflammatory diseases such as MS. It is produced by monocytes / macrophages and microglial cells and can exist in soluble or membrane form.the investigators of our clinical department were the first to describe the pro-inflammatory role of TWEAK in MS. Indeed, we have demonstrated in an animal model of MS that the inhibition of TWEAK makes it possible to reduce the severity of the disease. Our recent work (manuscript submitted for publication) has also shown results from a series of 28 patients with MS suggesting that the serum TWEAK assay may be an early marker of thrust occurrence. the investigators propose to study the concentration variations of the serum soluble form of cytokine TWEAK during the first year of MS and to analyze their correlation with the occurrence of an inflammatory disease outbreak. the investigators will perform a prospective study in which 50 patients with MS in the isolated clinical syndrome stage will be included over a 12-month period. Mental Cerebral MRIs will be performed for each patient at baseline (T0), month 6, and month 12. Serum dosages of TWEAK will be performed each month for each patient for one year. Patients will also be treated with soluble TNF, the leader in the TNF family of ligands, anti-TWEAK antibodies (which may interfere with the activity and dosage of TWEAK) as well as C-reactive Protein C ( search for intercurrent infectious episode). These dosages will be correlated with the clinical evolution (appearance or not of an inflammatory flare) as well as the data of the imagery (number of lesions raised or not by the gadolinium).

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 45 years
* the first inflammatory and demyelinating episode of the central nervous system affecting the optic nerve, the spinal cord
* No neurological antecedent demyelinating
* differential differential diagnosis at inclusion on the basis of clinical examination and biological examinations
* respect of the revised diagnostic criteria of Mac Donald 2010
* handicap degree between 0 and 5 at the time of diagnosis

Exclusion Criteria:

* pregnant woman

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
The serum concentration of soluble TWEAK | 1 year
  We will then compare the soluble TWEAK concentrations observed in patients with anti-TWEAK antibodies and in patients without anti-TWEAK antibodies. We will study the correlation between the concentrations of soluble TWEAK and those of soluble TNF.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Olivier ARNAUD, Study Director — Assistance Publique des Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France